CLINICAL TRIAL: NCT04781556
Title: Impact of Osteoporotic Fractures on Work: Data From a Fracture Liaisons Service
Acronym: OPTIWORK
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: OPTIWORK
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Osteoporotic Fractures
Keywords: osteoporotic fractures; work; quality of life
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — All patients treated between 01/01/2017 and 12/31/2018 in the Fracture sector will be screened through the computerized medical file. For patients who meet all the eligibility criteria, the information note, study questionnaire and a stamped envelope will be sent to them by post. Without feedback from him within 30 days of this submission, the patient is considered not to have objected to the study. The patient's information as well as his non-objection will be recorded in his medical file.

SUMMARY:
Osteoporosis is a bone disease characterized by a decrease in bone density with deterioration of the micro-architecture and the appearance of bone fragility, responsible for an increased risk of fractures. The most common osteoporotic fractures are spinal, wrist and femoral neck fractures. Osteoporosis affects 22.7% of women and 6.9% of men in France. Each year, around 8.9 million fragility fractures are identified worldwide, with an incidence in France in 2017 of 382,000 patients in France in 2017.

The economic impact, the functional consequences and the quality of life of patients with osteoporosis, fracture or not, have been widely described in the literature in recent years. There is indeed a great alteration in the mobility, functional capacities and overall quality of life of these patients, measured by composite scores such as Short Form-36 (SF-36), EuroQol 5 Dimensions (EQ-5D) , the Health-related quality of life (HRQoL), or more specifically for osteoporosis, osteoporososis quality of life questionnaire (OQLQ) or its shortened version OLQ, the osteoporosis assessment questionnaire (OPAQ), the Quality of life questionnaire of the European Foundation for Osteoporosis (QUALEFFO) (specific for vertebral fractures), etc.

However, few studies have focused on the repercussions of osteoporotic fractures at work, because this pathology affects more elderly subjects (> 65 years old) and therefore retirees.

DETAILED DESCRIPTION:
New osteoporosis management programs have emerged in recent years, in order to improve the management of this pathology by linking the specialties concerned. Among them, La Filière Fracture (in Anglo-Saxon: Fractures Liaisons Services: FLS) of the Paris Saint-Joseph Hospital Group (GHPSJ), created in 2015, aims to follow up patients consulting the GHPSJ for an osteoporotic fracture of spinal location. , the upper end of the femur or the lower end of the radius.

Since the creation of the sector, 2,486 patients have been recruited; it was found that in 529 of these patients (or 21.3%), the osteoporotic fracture occurred at an age of less than 65 years.

The impact on the work of an osteoporotic fracture has been little studied in the literature: a study focused specifically on fractures of the upper extremity of the femur, and found, in 291 patients under 65 years recruited between 2009 and 2013, a 65% return to work rate at 12 months, or around a third of patients who have not returned to professional activity at one year. A study published in 2016 assessed return to work delay and factors associated with return to work in 275 patients with fragility fractures in Canada; 88% had returned to work with an average absenteeism period of 20.5 days. The average duration of presenteeism (presence at work but with reduced productivity due to the fracture) was 2.9 hours in 4 weeks. Another Japanese study found a risk ratio of 4 (p <0.001) to greater absenteeism in patients with several osteoporotic fractures, with no difference found in terms of productivity at work compared to patients with a history of a single fracture or without history of osteoporotic fracture. The female sex, the need for surgical management, the existence of work with the need to carry heavy loads were associated with a prolonged return to work time.

The objective here is to assess the occupational impact of osteoporotic fractures occurring in active patients under 65 years of age, and to look for factors predicting a return to work within 3 months after the fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 at the time of the fracture
* French-speaking patient
* Patients treated in the Fracture Line between January 1, 2017 and December 31, 2018 for osteoporotic fracture
* Professionally active patients at the time of the fracture

Exclusion Criteria:

* Refusal to participate in the study
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated between 01/01/2017 and 31/12/2018 in the Fracture sector will be screened through the computerized medical file
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
To assess the consequences of osteoporotic fractures on the rate of return to work at 3 months of active patients under 65 years of age | Month 3
  Rate of patients returning to work 3 months after fracture

SECONDARY OUTCOMES:
To assess the consequences of osteoporotic fractures on the average return to work time of active patients under 65 years of age. | Day 1
  Average time to return to work
Evaluate the consequences of osteoporotic fractures on quality of life in active patients under 65 | Month 3
  Quality of life Short Form - 36 (SF36 scale)
Define the predictive factors for not returning to work. | Day 1
  Correlation (uni and multivariate regression) between returning to work or not and certain parameters such as personal and professional characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Agnès PORTIER, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France